CLINICAL TRIAL: NCT06757309
Title: Randomized Study to Evaluate the Impact of Dietary Optimization on Metabolic Profile, Immunoactivation and Cardiovascular Risk in HIV Population on ART
Brief Title: Impact of Mediterranean Diet in Cardiovascular Risk Among People With HIV
Acronym: VIHMED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022/10496/I
Record Dates: First submitted 2024-12-22; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-07

CONDITIONS: HIV Infection; Inflammation; Cardiovascular Risk; Mediterranean Diet
Keywords: HIV; Inflammation; Coronary Artery
MeSH Terms: conditions — HIV Infections; Inflammation | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care arm will be the management as currently is provided. It provides participants with general dietary advice through informational leaflets. No personalized counseling or follow-up sessions are included. Participants continue their usual diet, receiving only baseline and routine assessments without additional support to modify their dietary habits or improve adherence to healthier eating patterns.
- Intervention (Experimental): Intervention consists in personalized counseling to adopt the Mediterranean diet, focusing on whole foods, healthy fats, and lean proteins. Participants receive tailored meal plans, educational materials, and practical tips. Follow-up sessions at weeks 4 and 12 offer support, progress reviews, and goal-setting to ensure adherence and improved health outcomes.
  Interventions: Behavioral: Mediterranean Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — Intervention consists in personalized counseling to adopt the Mediterranean diet, focusing on whole foods, healthy fats, and lean proteins. Participants receive tailored meal plans, educational materials, and practical tips. Follow-up sessions at weeks 4 and 12 offer support, progress reviews, and goal-setting to ensure adherence and improved health outcomes
  Arms: Intervention

SUMMARY:
This study (VIHMET) aims to explore how dietary changes, specifically the adoption of a Mediterranean diet, can improve health outcomes in people living with HIV (PLWH) who are on antiretroviral therapy (ART). PLWH often experience chronic inflammation, metabolic disturbances, and elevated cardiovascular risk due to the virus, immune activation, and ART-related side effects. By examining dietary interventions, this study seeks strategies to reduce these risks and enhance quality of life.

The VIHMET study is a randomized clinical trial involving 64 participants at Hospital del Mar, Barcelona, randomized into control and intervention groups (1:2 ratio). The intervention group will receive personalized nutritional counseling to improve adherence to the Mediterranean diet, focusing on food selection and meal preparation. The control group will follow standard dietary recommendations. Assessments will occur at baseline, week 24, and week 48.

Key health indicators include lipid profiles, markers of inflammation, immune activation, and cardiovascular health, assessed through non-invasive techniques like arterial stiffness and subclinical atherosclerosis measurements. Participants will complete questionnaires on diet adherence, physical activity, and quality of life, alongside anthropometric evaluations.

Eligible participants are adults with HIV, undetectable viral loads for 12+ months, and elevated LDL cholesterol with low Mediterranean diet adherence. Exclusion criteria include lipid-lowering drugs, chronic anti-inflammatory therapy, or other active inflammatory/metabolic conditions.

This study aims to improve lipid levels, reduce inflammation, decrease arterial stiffness, and assess diet adherence's impact on quality of life and subclinical atherosclerosis. Results may inform dietary recommendations to reduce cardiovascular risks and enhance holistic care for PLWH.

DETAILED DESCRIPTION:
The VIHMET study aims to investigate the role of dietary optimization, specifically adopting a Mediterranean diet, in improving metabolic health, reducing immune activation, and mitigating cardiovascular risks in people living with HIV (PLWH) who are on antiretroviral therapy (ART). PLWH face unique challenges, including chronic immune activation and increased inflammation, which contribute to accelerated aging, metabolic complications, and a higher prevalence of cardiovascular disease (CVD) compared to the general population. This study hypothesizes that dietary interventions may reduce these risks, leading to better overall health outcomes.

Study Design

This randomized, prospective, open-label interventional study will recruit 64 participants from the HIV outpatient clinic at Hospital del Mar in Barcelona. Participants will be randomized into two groups: an intervention group and a control group ( 1 SoC:2 intervention ratio). The intervention group will receive personalized counseling to improve adherence to the Mediterranean diet, while the control group will receive general dietary recommendations. Each participant will be followed for 48 weeks, with clinical and laboratory evaluations conducted at baseline, week 24, and week 48.

Study Objectives

Primary Objectives:

To evaluate changes in lipid profiles (total cholesterol, LDL, HDL, and triglycerides) at weeks 24 and 48.

To assess reductions in immune activation markers and inflammatory cytokines, such as IL-6, TNF-alpha, and sCD14.

To measure improvements in arterial stiffness using pulse wave velocity (PWV) as an indicator of subclinical CVD.

To assess the impact of the intervention on adherence to the Mediterranean diet using the MEDAS score.

Secondary Objectives:

To evaluate changes in quality of life using the EQ-5D questionnaire. To analyze changes in body composition, including BMI, waist circumference, and weight.

To assess reductions in TMAO (trimethylamine-N-oxide), a biomarker linked to CVD risk.

To investigate the presence and composition of coronary atherosclerosis using non-invasive coronary CT angiography (CCTA).

Participant Eligibility

Inclusion Criteria:

Adults aged 18 years or older. Confirmed HIV diagnosis. On stable ART with an undetectable viral load for at least 12 months. LDL cholesterol >140 mg/dL. Mediterranean Diet Adherence Screener (MEDAS) score <9, indicating low adherence.

Exclusion Criteria:

Use of lipid-lowering medications or chronic anti-inflammatory drugs. Active hepatitis B or C or other chronic inflammatory conditions. Familial hypercholesterolemia. Uncontrolled hypothyroidism or diabetes mellitus. Inability to provide informed consent.

Interventions Ratio: 1 SoC : 2 intervention

Intervention Group: Participants in the intervention group will undergo tailored nutritional counseling focusing on the Mediterranean diet. Key components include:

Education on food selection and preparation, emphasizing fruits, vegetables, whole grains, olive oil, nuts, and fish.

Guidance on reducing saturated fats and sugars. Development of individualized meal plans considering dietary habits and socioeconomic status.

Scheduled virtual follow-ups at weeks 4 and 12 to review adherence and address challenges.

Control Group: Participants will receive general dietary advice provided through standard informational leaflets. No individualized or follow-up counseling will be provided.

Outcome Measures

Primary Outcomes:

Changes in lipid profiles (total cholesterol, LDL, HDL, and triglycerides) at week 24 and 48 respect to baseline Reductions in inflammatory and immune activation markers (IL-6, TNF-alpha, sCD163, and sCD14) at week 24 and 48 respect to baseline Improvements in arterial stiffness as measured by PWV at week 24 and 48 respect to baseline

Secondary Outcomes:

Improvements in MEDAS scores, indicating better adherence to the Mediterranean diet at week 24 and 48 respect to baseline Changes in TMAO levels, reflecting reduced CVD risk at week 24 and 48 respect to baseline Alterations in quality of life (EQ-5D scores) at week 24 and 48 respect to baseline Presence and composition of coronary plaques using CCTA.

Procedures and Assessments

Participants will attend clinical visits at baseline, week 24, and week 48. The following assessments will be conducted:

Clinical Data Collection:

Medical history, HIV-related parameters, and medication use. Anthropometric Measurements: BMI, waist circumference, and weight. Dietary Adherence: MEDAS score and food frequency questionnaires. Laboratory Tests: Lipid profiles, inflammatory markers, immune activation biomarkers, and TMAO levels.

Imaging: Pulse wave velocity and CCTA to evaluate arterial health and coronary plaque burden.The study aims to demonstrate the benefits of dietary interventions in reducing CVD and metabolic risks, offering a holistic approach to HIV care that integrates nutritional counseling for long-term health improvements.

Statistical Analysis

Data will be analyzed using appropriate statistical methods. Continuous variables will be expressed as means and standard deviations, while categorical variables will be reported as frequencies. Comparisons between groups will be performed using t-tests or non-parametric equivalents, depending on data distribution. Multivariate regression models will assess the independent effects of dietary intervention on primary and secondary outcomes. All analyses will be conducted using Stata software, and a p-value <0.05 will be considered statistically significant. A sample size of 60 participants (40 in the intervention group and 20 in the control group) provides adequate power to detect clinically significant changes in LDL cholesterol and other outcomes.

Ethical Considerations

The study adheres to the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. All participants will provide written informed consent, and data confidentiality will be maintained according to GDPR standards. Participants will not receive financial compensation but will benefit from detailed health assessments and personalized dietary guidance.

Expected Impact

This study is expected to provide valuable insights into the role of dietary optimization in reducing cardiovascular and metabolic risks in PLWH. By addressing chronic inflammation, lipid disturbances, and immune activation, the findings could inform new strategies for integrating dietary counseling into HIV care. Such an approach emphasizes a holistic perspective, considering not only virological control but also long-term health and quality of life. The VIHMET study could represent a significant step forward in personalized care for PLWH, with potential applications in broader chronic disease management.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Confirmed diagnosis of HIV infection.
* On stable antiretroviral therapy (ART) with an undetectable viral load for at least 12 months.
* LDL cholesterol levels >140 mg/dL.
* Low adherence to the Mediterranean diet, defined by a MEDAS score <9.
* Must be able to swallow tablets
* Willingness and ability to provide informed consent.

Exclusion Criteria:

* Use of lipid-lowering medications.
* Chronic use of anti-inflammatory drugs.
* Active hepatitis B or hepatitis C infection.
* Other chronic inflammatory conditions (e.g., autoimmune diseases).
* Familial hypercholesterolemia.
* Uncontrolled metabolic conditions, such as hypothyroidism or diabetes mellitus.
* Pregnancy or breastfeeding.
* Cognitive or psychological conditions impairing the ability to comply with the study protocol.
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in LDL profile between groups | 24 weeks
  Difference in the mean change (mg/dL) in LDL cholesterol between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values.
Changes in HDL cholesterol | week 24 respec to baseline
  Difference in the mean change (mg/dL) in HDL cholesterol between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values.
Changes in body mass index | 24 weeks
  Difference in the mean change in body Mass Index between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values.
Changes in very low density lipoprotein by spectral MRI | 24 weeks
  Difference in the mean change in very low lipoprotein between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values measured by spectral MRI

SECONDARY OUTCOMES:
Changes in CD38+CD4+T-cell | 24 weeks
  Difference in the mean percentage change in CD38+CD4+ T-cell levels between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values, as measured by flow cytometry.
Changes in CD38+CD8+T-cell | 24 weeks
  Difference in the mean percentage change in CD38+CD8+T-cell levels between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values, as measured by flow cytometry.
change in Exhaustion CD4 T-cells | 24 weeks
  Difference in the mean percentage change in PD1+CD4+T-cells levels between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values, as measured by flow cytometry.
Changes in PD1+CD8+T-cells | week 24
  Difference in the mean percentage change in PD1+CD8+T-cells levels between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values, as measured by flow cytometry.
Change in Pulse wave velocity | week 24
  Difference in the mean percentage change in the Pulse Wave Velocity between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values.
Change in Pulse wave velocity 48w | Week 48
  Difference in the mean percentage change in the Pulse Wave Velocity between the intervention group and the standard of care (SoC) group at week 48, relative to baseline values.
Changes in MEDAS score | 24 week
  Difference in the mean percentage change in the MEDAS score between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values.
changes in MEDAS score at week 48 | Week 48
  Difference in the mean percentage change in the MEDAS score between the intervention group and the standard of care (SoC) group at week 48, relative to baseline values.
Changes Quality of life measured by EQ-5D-3L at week 24 | week 24
  Difference in the mean percentage change in score of Quality of life measured by EQ-5D-3L between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values.
Changes Quality of life measured by EQ-5D-3L at week 48 | 48 weeks
  Difference in the mean percentage change in score of Quality of life measured by EQ-5D-3L between the intervention group and the standard of care (SoC) group at week 48, relative to baseline values.
Changes in Calcium Score | week 24
  Difference in the mean percentage change in Calcium score Agatston between the intervention group and the standard of care (SoC) group at week 24, relative to baseline values, measured by angio-CT coronary scan.
Changes in Calcium Score | 48 weeks
  Difference in the mean percentage change in Calcium score Agatston between the intervention group and the standard of care (SoC) group at week 48,relative to baseline values, measured by angio-CT coronary scan.
Changes in Lipid core of the coronary plaque by week 24 | Week 24
  Difference in the mean percentage change in the lipid proportion of the coronary plaque between the intervention group and the standard of care (SoC) group at week 24 ,relative to baseline values, measured by angio-CT coronary scan.
Changes in the lipid core of the coronary plaque by week 48 | 48 weeks
  Difference in the mean percentage change in the lipid proportion of the coronary plaque between the intervention group and the standard of care (SoC) group at week 48 ,relative to baseline values, measured by angio-CT coronary scan.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Güerri-Fernández, M.D. Ph.D., Study Chair — Hospital del Mar; Juan Jose Chillarón-Jordan, M.D. Ph.D., Study Chair — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on demand upon reasonable request, in compliance with ethical guidelines and applicable data protection regulations.

DOCUMENTS (2):
  • Study Protocol (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT06757309/Prot_000.pdf
  • Informed Consent Form (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT06757309/ICF_001.pdf